CLINICAL TRIAL: NCT02845206
Title: Randomised Controlled Trial of Patient Specific Instrumentation vs Standard Instrumentation in Total Knee Arthroplasty
Brief Title: Bespoke vs Standard Instrumentation in TKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 15/SS/0058
Record Dates: First submitted 2016-03-21; First posted 2016-07-27 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Replacement; Patient Specific Instrumentation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Specific Cutting Blocks (Experimental): For the bespoke individualised cutting blocks to be manufactured, the patients will undergo a preoperative CT scan under a set protocol. The CT radiation dose will be considerably less than a conventional diagnostic CT scan.
  Interventions: Procedure: Patient specific cutting blocks
- Conventional Cutting Blocks (Active Comparator): The patients in this arm will be operated on using conventional instruments.
  Interventions: Procedure: Conventional cutting blocks

INTERVENTIONS:
Procedure: Patient specific cutting blocks — 'MyKnee' Instrumentation
  Arms: Patient Specific Cutting Blocks
Procedure: Conventional cutting blocks — Standard Instrumentation
  Arms: Conventional Cutting Blocks

SUMMARY:
Total knee replacement (TKR) is an established treatment for knee osteoarthritis and leads to a satisfactory outcome in over 75% of patients. The pain and function after TKR can be dependent on the accuracy of initial implantation, as deviation of more than 3 degrees from the normal alignment of the limb can lead to abnormal stresses on the implant and accelerated failure. Patient specific cutting blocks may result in a more individualised implant placement, improved pain and function following surgery, and a long-lasting implant.

This trial is designed to investigate if there is any benefit to bespoke instrumentation in terms of pain and function to the patient, and an economic benefit to the NHS.

DETAILED DESCRIPTION:
Total knee replacement (TKR) is an established treatment for 'wear and tear' arthritis and leads to a satisfactory outcome in over 75% of patients. However, this means that up to 25% of patients are not entirely satisfied with their TKR. The longevity and stability of a TKR is greatly dependent on the accuracy of the initial surgery. Deviation of more than 3 degrees from the normal axis can lead to abnormal stresses causing the implants to fail. 'Patient specific' technology involves preoperative computer assessment of the patients' knee and allows for a 'patient specific' cutting block to be manufactured. This will allow for individual bony cuts specific to the patients own anatomy.

'Patient specific' implants and cutting blocks may allow a more optimal implant positioning and are implanted without the need for instrumentation of the femoral medullary canal (thigh), so lower blood loss may result. This could result in improved early range of movement and decreased pain following surgery. The total knee replacement used in this study will be the GMKSphere (Medacta International) TKR. It has a specific design which more closely resembles a natural unreplaced knee than any other knee replacement. It may help address the phenomenon of 'mid flexion instability', which is where the patient perceives their replaced knee to be unsteady on stairs and slopes.

Patient specific technology may also result in a cost saving, as it potentially reduces the number of sterilised trays required during the surgery.

This study will allow for comparison in knee function and patient outcomes between patients who have undergone their TKR with patient specific cutting blocks compared to conventional cutting blocks. The scans obtained following the surgery could lead to world leading methodology for the assessment of knee replacements and would set a blue print for the evaluation of other knee implants in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis ('wear and tear') of the knee which is sufficiently symptomatic to require knee arthroplasty as assessed by their consultant orthopaedic surgeon

Exclusion Criteria:

* Patients with inflammatory arthropathy, patients requiring bone augmentation, ligament incompetence, values deformity > 5 degrees

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Limb alignment | 1 years
  Measured in degrees from Hip-Knee-Ankle radiographs from centre of femoral head to midpoint of the ankle

SECONDARY OUTCOMES:
Difference between baseline pre-op and one year post-op change in gait measured using a bespoke clinic-appropriate motion analysis system. | 1 year
  Knee range of motion, strength and gait analysis assessments will be carried out on a bespoke clinic-appropriate motion analysis system. This system consists of 8 Vicon B10 Bonita cameras (Vicon Systems, Oxford) which immediately surround a self-paced N-Mill treadmill (Motekforce Link, Amsterdam).
Difference in patient reported knee pain level as measured by Oxford Knee Score between baseline and one year and also between study groups. | 1 year
  Validated patient reported knee pain questionnaires as measured by Oxford Knee Score (out of 48 points) pre-operation and at one year post-operation. Difference between baseline and one year scores for each patient and also analysed between groups (patient specific cutting blocks compared to conventional cutting blocks).
Difference in patient reported knee function between baseline and one year and also between study groups. | 1 year
  Validated patient reported knee function questionnaires as measured by EQ-5D pre-operation and at one year post-operation. Difference between baseline and one year scores for each patient and also analysed between groups (patient specific cutting blocks compared to conventional cutting blocks).
Difference in patient reported quality of life questionnaires between baseline and one year and also between study groups. | 1 year
  Validated quality of life questionnaires as measured by SF-12 score pre-operation and at one year post-operation. Difference between baseline and one year scores for each patient and also analysed between groups (patient specific cutting blocks compared to conventional cutting blocks).
Healthcare cost | 1 year
  Healthcare cost measured in pounds sterling (GBP). Total cost of performing knee replacement using conventional cutting blocks compared to using bespoke cutting blocks and disposable instrumentation. The measurable contributors to the costs of healthcare include operating time (minutes), number of instrument trays requiring sterilisation (number of trays), length of hospital stay (days), patient transfusion requirement (number of units of packed cells required), cost of bespoke disposable instrumentation (GBP).

CONTACTS AND LOCATIONS:
Overall Officials: Leela C Biant, FRCSEd(Tr&Orth) MSres MFSTEd, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data available to bone fide researchers at the end of the study